CLINICAL TRIAL: NCT01438879
Title: Molecular Methods in the Etiological Diagnostics of Acute Central Nervous System Infections: Lymphocytic Herpesviruses and PCR
Brief Title: Lymphocytic Herpesviruses and Cerebrospinal Fluid Polymerase Chain Reaction (PCR)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PaijatHame Central Hospital (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Laura Kupila, Specialist in neurology, MD PhD, PaijatHame Central Hospital
Other Study IDs: R11077
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Central Nervous System Infection
Keywords: CSF; PCR; lymphocytic herpesvirus; CNS
MeSH Terms: conditions — Central Nervous System Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF white cells + CSF supernatant, Blood white cells and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pleocytosis group: 40 patients with clinical signs of CNS infection and having CSF pleocytosis.
- non-pleocytosis group: 20 patients not having CNS infection clinically and not having CSF pleocytosis.

SUMMARY:
Enterovirus and herpes simplex viruses 1 and 2 are the main causative agents of central nervous system infections.

Instead, the role of lymphocytic herpesviruses in the etiology of central nervous system (CNS) infections is not clear, even if there is the positive cerebrospinal fluid (CSF) polymerase chain reaction (PCR)-result for the virus.

The aim of this study is to evaluate the presence of DNA from lymphocytic herpesviruses in the CSF obtained from the immunocompetent patients with CSF pleocytosis and from the patients with normal CSF leukocyte count.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent patients with clinical symptoms and signs of central nervous system infections and CSF pleocytosis (pleocytosis group)
* Immunocompetent patients without suspicion of CNS infection and no CSF pleocytosis (non-pleocytosis group)

Exclusion Criteria:

* Suspicion of CNS-infection, eg. encephalitis, but no CSF leukocytosis (pleocytosis group)
* Patients without symptoms of CNS infection, but who has CSF pleocytosis of unknown origin (non-pleocytosis group)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of the district of Paijat-Hame (200 000 inhabitants).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laura MA Kupila, Principal Investigator — PaijatHame Central Hospital
Locations (1):
- PaijatHame Central Hospital, Lahti, Finland